CLINICAL TRIAL: NCT04515693
Title: Exploring Psychometric Properties of a New Version of the 6MWT in the Acute Stroke Population
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID there were limitations is performing study activities and it was decided to terminate the study.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Megan C. Eikenberry, P.T., D.P.T., Assistant Professor of Physical Therapy, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-010067
Record Dates: First submitted 2020-08-14; First posted 2020-08-17 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Maximal Assist group (Experimental): Subjects with acute stroke who ambulate with Maximal assistance of 1.
  Interventions: Other: 6 Minutes Walking Test
- Moderate Assist group (Experimental): Subjects with acute stroke who ambulate with Moderate assistance of 1.
  Interventions: Other: 6 Minutes Walking Test
- Minimal Assist group (Experimental): Subjects with acute stroke who ambulate with Minimal assistance of 1.
  Interventions: Other: 6 Minutes Walking Test
- Supervision/Modified Independence/Independence (Experimental): Subjects who walk without physical assistance of a helper.
  Interventions: Other: 6 Minutes Walking Test

INTERVENTIONS:
Other: 6 Minutes Walking Test — A walkway of 12 meters will be marked with one cone at each end. The patient will be instructed to walk back and forth as many times as possible in six minutes.

SUMMARY:
The purpose of this study is to assess inter- and intra-rater reliability of the 6MWT in people with acute stroke who require various levels of assistance with walking.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Primary diagnosis of an acute or hemorrhagic stroke
* Admitted into the acute or acute rehab setting and is appropriate for physical therapy services.
* Can ambulate with 1 person assistance and a device as needed, with no more than maximal assistance required. The patient must be able to independently advance the lower extremity forward, but can receive maximal assistance for blocking, bracing or postural control during ambulation.
* Can stand and/or ambulate for at least 6 minutes

Exclusion Criteria:

* Hemodynamically unstable
* Unstable medical co-morbidities such as: active bleeding, recurring seizures, uncontrolled hypertension (permissive HTN orders ok)
* Patients with bilateral acute stroke
* Patients who are unable to follow 1 step commands as determined by the screening physiatrist
* Orthopedic co-morbidities that place a weight-bearing restriction on the lower extremities such as acute fracture, joint replacement, or other musculoskeletal injury
* Any other condition that would limit a patient's ability to remain in a standing position with assistance for 6 minutes at a time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
6 Minute walk test | 8 minutes (2 minutes for set-up, 6 minutes to execute)
  walking endurance assessment measured in meters of total distance completed over 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Karstetter, PT, DPT, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials